CLINICAL TRIAL: NCT05998499
Title: HIV-Infected Latin American Asylum Seekers in Europe: Insights From the EuroLatin HIV Cohort (ELHC)
Brief Title: HIV-Infected Latin American Asylum Seekers in Europe: Insights From the EuroLatin HIV Cohort
Acronym: ELHC
Status: Completed | Type: Observational
Sponsor: Hospital Universitario Infanta Leonor (Other)
Responsible Party: Principal Investigator, Pablo Ryan, Principal Investigator, Hospital Universitario Infanta Leonor
Other Study IDs: HUIL_MI_VIH01
Record Dates: First submitted 2023-08-10; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: HIV-1-infection; Sexually Transmitted Diseases
Keywords: Asylum Seekers; Migration; Europe; Latin America
MeSH Terms: conditions — Sexually Transmitted Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- EuroLatin HIV Cohort (ELHC): Cohort of Latin American migrants living with HIV who were seeking international protection in Spain (Europe)
  Interventions: Other: Description

INTERVENTIONS:
Other: Description — This study aimed to understand the situation of Latin American HIV-positive migrants seeking asylum in Spain and identify the challenges they encounter in getting HIV treatment. The main result measured was the proportion of participants with an HIV-1 RNA level of 50 copies/mL or higher at their first clinic visit

SUMMARY:
This is a longitudinal observational study conducted in Europe that describes migrants infected with HIV from Latin America who come to Europe with the intention of seeking asylum or international protection. The aim of the study is to identify the barriers this population faces in accessing the healthcare system and to assess disease control

DETAILED DESCRIPTION:
Study Design and Setting This observational study was conducted between 2022 and 2023 in Madrid, Spain. Participants were recruited at the HIV outpatient clinic of Infanta Leonor University Hospital (HUIL) for the study and were monitored for a period of 6 months from their enrollment in the study.

Participant Recruitment Participants were primarily identified and referred by various non-governmental organizations (NGOs) working with migrants living with HIV. These NGOs, which included gTt-VIH, Apoyo Positivo, Cogam, Acción Triangulo, Kif-Kif, Salud Entre Culturas, and the Spanish Red Cross, played an essential role by establishing a crucial link and provided a vital bridge, facilitating the patients' integration into the healthcare system through an unconventional circuit.

Medical Evaluation In the HIV unit, assessments were conducted by experienced infectious disease specialists and a unit-specific nurse. The care protocol comprised a meticulous collection of medical history, an exhaustive physical examination, along with a series of tests. Furthermore, appointments were scheduled for a one-month and six-month follow-up to ensure continuous care and monitor the effectiveness of the treatment regimen.

Social and Psychological Evaluation An experienced social worker with a background in vulnerable populations was hired to perform a social assessment. Six months post the initial hospital visit, the social worker re-established contact with the patients to reassess their social circumstances and their continued engagement with the HIV consultation services.

Ethical Considerations This study adhered to the ethical principles outlined in the Declaration of Helsinki and received the necessary approvals from the ethics committee at Infanta Leonor Hospital. Informed consent was provided by every participant.

Data collection In this study, the REDCap application was utilized for the collection of data. The database was stored in a secure server, and only researchers and health personnel of the project had access to it.

ELIGIBILITY:
Inclusion Criteria:

* Latin American migrants infected with HIV who arrive in Spain with the intent to seek international protection and who lack access to healthcare.

Exclusion Criteria:

* Those who do not give their consent

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Latin American migrants infected with HIV
Sampling Method: Non-Probability Sample
Enrollment: 631 (Actual)
Dates: Start 2022-01-30 (Actual); Primary Completion 2023-04-30 (Actual); Study Completion 2023-07-15 (Actual)

PRIMARY OUTCOMES:
HIV viral control | At inclusion
  Number of participants with plasma HIV-1 RNA level of more than 50 copies per mL

SECONDARY OUTCOMES:
Resistance Pattern | At inclusion
  Number of participants with Drug Resistance
Sexually transmited infections | At inclusion
  Number of participants with sexually transmited infections
Number and Type of Barriers to Accessing Healthcare | At inclusion
  The outcome will assess the number and type of barriers faced by study participants when trying to access healthcare, based on the presence of any of the following barriers: administrative, geographical, financial, cultural, lack of knowledge, stigma, and organizational.
HIV viral control at 6 months | 6 months
  Number of participants with plasma HIV-1 RNA level of more than 50 copies per mL
Retention in care | 6 months
  Number of participants who maintain retention to healthcare

CONTACTS AND LOCATIONS:
Overall Officials: Pablo Ryan Murua, MD, PhD, Principal Investigator — Hospital Universitario Infanta Leonor
Locations (1):
- Hospital Universitario Infanta Leonor, Madrid, Spain

IPD SHARING:
Plan to Share IPD: Yes
IPD that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: December, 2024
Access Criteria: IP email